CLINICAL TRIAL: NCT06516458
Title: Development of Camera Based Gait Deviation Index for Persons With Multiple Sclerosis
Brief Title: Development of Camera Based Gait Quality Measure for Persons With Multiple Sclerosis
Acronym: MS-GDI
Status: Recruiting | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Milap Sandhu, Principal Investigator, Shirley Ryan AbilityLab
Other Study IDs: STU00221990
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Secondary Progressive; Multiple Sclerosis Relapse; Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Gait quality observation
  Interventions: Diagnostic Test: Camera Based Kinematic Analysis

INTERVENTIONS:
Diagnostic Test: Camera Based Kinematic Analysis — Observational Study using Camera Based, Marker Less Kinematic Analysis of gait quality of persons with Multiple Sclerosis
  Other Names: OpenCap

SUMMARY:
The purpose of this study is to develop a measurement of walking quality, called Gait Deviation Index (GDI) for people with Multiple Sclerosis (MS).

DETAILED DESCRIPTION:
In rehabilitation in general, in order to track patients' progress and provide next steps, there is a need for easily obtainable, understandable, and objective measures of ability. Currently, there is no measure that clinicians can utilize to determine walking quality. While Gait Deviation Index has been validated and can reliably be used in adults who experienced a Spinal Cord Injury, it has not yet been validated in people with MS. After the MS-specific GDI is developed from this study, therapists and clinicians will be able use it as a reliable progress measure. Which may lead to the delivery of more effective therapy for patients with MS.

Here we plan to measure body position with camera based tracking during your gait cycle.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of relapsing form of MS (including relapsing-remitting MS and secondary progressive MS)
* Able to ambulate overground
* Relapse free for at least 1 month
* Age ≥18 and ≤ 75 years
* Participants using dalfampridine will be eligible if taking the same daily dose for at least 2 months prior to screening

Exclusion criteria:

- Orthopedic injuries, fractures, surgeries or other conditions affecting locomotor function or weight bearing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with multiple sclerosis who can ambulate overground
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Kinematics of the gait cycle | at the time of session
  Joint position of lower limbs during a single cycle of gait

SECONDARY OUTCOMES:
6 minute walk test | at the time of session
  you will be instructed to walk as quickly and safely as you can while being timed for 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Milap Sandhu, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Share overall data set